CLINICAL TRIAL: NCT02661828
Title: A Comparison of Two Antidepressant Tapering Regimens
Brief Title: Tapering Off Antidepressants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Boadie W. Dunlop, Boadie W. Dunlop, MD, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00084849
Record Dates: First submitted 2016-01-20; First posted 2016-01-25 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-01

CONDITIONS: Major Depressive Disorder; Anxiety Disorder; Obsessive Compulsive Disorder; Post-Traumatic Stress Disorder
Keywords: Tapering Antidepressant Regimen; Antidepressant Discontinuation Syndrome
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taper A Regimen (Active Comparator): Participants taking an antidepressant for at least four weeks and no longer wish to take the antidepressant medication will undergo a Two-Week Taper Regimen to discontinue their medication.
  Interventions: Other: Two-Week Antidepressant Taper Regimen
- Taper B Regimen (Active Comparator): Participants taking an antidepressant for at least four weeks and no longer wish to take the antidepressant medication will undergo a One-Week Taper Regimen to discontinue their medication.
  Interventions: Other: One-Week Antidepressant Taper Regimen

INTERVENTIONS:
Other: Two-Week Antidepressant Taper Regimen — Days 1-7: 50% of baseline antidepressant dose taken; Days 8-14: 25% of baseline antidepressant dose taken; Day 15: Stop antidepressant.
  Arms: Taper A Regimen
Other: One-Week Antidepressant Taper Regimen — Days 1-3: 50% of baseline antidepressant dose taken; Days 4-7: 25% of baseline antidepressant dose taken; Day 8: Stop antidepressant.
  Arms: Taper B Regimen

SUMMARY:
The purpose of this study is to compare two ways to stop taking an antidepressant medication and determine whether a faster or slower taper is better tolerated.

DETAILED DESCRIPTION:
As abrupt cessation of antidepressant medication can cause distressing symptoms (including and not limited to worsened mood, irritability/agitation, anxiety, dizziness, confusion, and headache), the aim of this study is to compare the tolerance of two tapering regimens with the hypothesis that tapering the antidepressant dose over the course of two weeks will yield less discontinuation symptoms than a one week taper regimen. Additionally, it is suspected that discontinuing medications that inhibit the serotonin transporter , such as selective serotonin reuptake inhibitors (SSRI) and serotonin norepinephrine reuptake inhibitors (SNRI) will have a greater difference in the frequency of discontinuation symptoms between the two and one-week tapering regimens versus antidepressants that don't inhibit serotonin transporter.

Demographic and clinical features will also be identified that may predict discontinuation symptoms with the hypothesis that patients on SSRIs and SNRIs may experience more discontinuation symptoms versus patients on non-SSRI/SNRI medications. Whether or not the treatment duration is positively associated with the number of discontinuation symptoms will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Currently taking an FDA-approved antidepressant for at least four weeks on the list of approved medications: SSRIs (citalopram, escitalopram, fluoxetine, fluvoxamine, paroxetine, sertraline, vilazodone or vortioxetine), SNRIs (desvenlafaxine, duloxetine, levomilnacipran, venlafaxine) and other classes (amitriptyline, bupropion, desipramine, doxepin, mirtazapine, nefazodone, nortriptyline, phenelzine, selegiline, or tranylcypromine). Clomipramine, a tricyclic antidepressant approved for the treatment of OCD, will also be included, but will be classed as an SSRI for this study because inhibition of the serotonin transporter is its primary therapeutic mechanism.
* No longer wish to take the antidepressant medication they are currently prescribed, due to one of the following reasons: 1) ineffective for symptoms; 2) intolerable side effect; 3) improvement of their illness for sufficient duration that it is clinically appropriate to consider tapering the medication.
* Primary psychiatric diagnosis of major depressive disorder, an anxiety disorder, OCD, or PTSD.
* Ability to read and understand English language.

Exclusion Criteria:

* Has met criteria at any time during their life for a primary psychotic disorder (e.g. schizophrenia), or dementia.
* Meets criteria for DSM-5-defined substance use disorder within three months of the screening visit.
* Currently taking two or more antidepressants.
* Presents with a clinically significant suicide risk, as assessed by a study physician.
* Presence of any unstable or central nervous system-related medical illness that would interfere with cognition or participation.
* Women who are currently pregnant or lactating, or plan to become pregnant during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-01; Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boadie Dunlop, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - 12 Executive Park Drive, 3rd floor, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from January 2016 through March 2017.
Pre-assignment Details: Of the two participants who signed consent, one subject began study participation for which data were collected.
Period: Overall Study
Arm/Group | Taper A Regimen | Taper B Regimen
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects entered the Taper B Regimen Arm/Group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Taper A Regimen | Taper B Regimen | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Full Range); unit: years] | 47 [47 to 47] |  | 47 [47 to 47]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 1 |  | 1
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Discontinuation Emergent Signs and Symptoms Scale (DESS) Scores
Description: To determine a change in the frequency of Discontinuation symptoms, the Discontinuation Emergent Signs and Symptoms Scale (DESS) will be administered by a trained clinician/rater to assess the frequency of discontinuation symptoms. The assessment has 43 items to evaluate discontinuation-emergent symptoms resulting from withdrawal from their antidepressant medication. Symptoms are rated on a scale of 1-5:
  1. New symptom
  2. Old symptom but worse
  3. Old symptom but improved
  4. Old symptom but unchanged
  5. Symptom not present
  Total score = sum of number of new symptoms and old (but worse) symptoms (score = 1) and old and unchanged symptom, absent, or old symptom but improved (score = 0); total possible range 0 to 43. Higher score = more symptoms.
Time Frame: Baseline (Post-Taper), Visit 4 (3 Weeks Post Baseline)
Measure: Number; unit: units on a scale
Arm/Group | Taper A Regimen
Number analyzed (Participants) | 1
units on a scale
  Baseline (Post-Taper) | 0
  Visit 4 | 6

2. Secondary Outcome: Physician Withdrawal Checklist (PWC-20) Scores
Description: To determine a change in the Intensity of Discontinuation symptoms, the Physician Withdrawal Checklist (PWC-20) will be administered by a trained clinician/rater to assess the intensity of discontinuation symptoms. The assessment has 20 items evaluated to detect withdrawal symptoms. Symptoms are rated on a scale of 0-3.
  0. Not present
  1. Mild
  2. Moderate
  3. Severe
  Total scores range from 0 to 60 with higher scores indicating more severe symptoms.
Time Frame: Baseline (Post-Taper), Visit 4 (3 Weeks Post Baseline)
Measure: Number; unit: units on a scale
Arm/Group | Taper A Regimen
Number analyzed (Participants) | 1
units on a scale
  Baseline (Post-Taper) | 15
  Visit 4 | 15

3. Secondary Outcome: Number of Participants Who Meet Criteria for Antidepressant Discontinuation Syndrome
Description: Antidepressant Discontinuation Syndrome is defined as greater than or equal to 4 new or worsened Discontinuation Emergent Signs and Symptoms Scale (DESS) symptoms at a visit during the study.
  Symptoms are rated on a scale of 1-5:
  1. New symptom
  2. Old symptom but worse
  3. Old symptom but improved
  4. Old symptom but unchanged
  5. Symptom not present
Time Frame: Duration of Study (Up to 14 Months)
Measure: Count of Participants; unit: Participants
Arm/Group | Taper A Regimen
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: No subjects entered the Taper B Regimen Arm/Group.
Arm/Group | Taper A Regimen | Taper B Regimen
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02661828/Prot_SAP_000.pdf